CLINICAL TRIAL: NCT01876368
Title: A Randomized 8-week Double-blind, Parallel-group, Active-controlled, Multicenter Study to Evaluate Efficacy and Safety of LCZ696 200 mg in Comparison With Olmesartan 20 mg in Essential Hypertensive Patients Not Responsive to Olmesartan
Brief Title: Efficacy and Safety of LCZ696 Compared to Olmesartan in Essential Hypertensive Patients Not Responsive to Olmesartan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2318; 2013-001783-36 (EudraCT Number)
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: hypertension,; LCZ696,; olmesartan
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; olmesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCZ696 200 mg (Experimental): Patients will be treated with one LCZ696 200 mg tablet and one placebo of olmesartan 20 mg capsule once daily for 8 weeks.
  Interventions: Drug: LCZ696; Drug: Placebo of LCZ696
- Olmesartan 20 mg (Active Comparator): Patients will be treated with one placebo of LCZ696 200 mg tablet and one olmesartan 20 mg capsule once daily for 8 weeks.
  Interventions: Drug: Olmesartan; Drug: Placebo of Olmesartan

INTERVENTIONS:
Drug: LCZ696
  Arms: LCZ696 200 mg
Drug: Olmesartan
  Arms: Olmesartan 20 mg
Drug: Placebo of LCZ696
  Arms: LCZ696 200 mg
Drug: Placebo of Olmesartan
  Arms: Olmesartan 20 mg

SUMMARY:
This study will assess the efficacy and safety of LCZ696 in comparison to olmesartan in essential hypertensive patients not adequately responsive to olmesartan

ELIGIBILITY:
Inclusion Criteria:

* patients with mild to moderate hypertension, untreated or currently taking antihypertensive therapy
* treated patients (using antihypertensive drugs within 4 weeks prior to first visit) must have an office msSBP ≥ 145 mmHg and < 180 mmHg after washout epoch and after 4 weeks run-in epoch
* untreated patients (either newly diagnosed or those patients with a history of hypertension but have not been taking any antihypertensive drugs for at least 4 weeks prior to first visit) must have an offcie msSBP ≥ 150 mmHg and < 180 mmHg at screening and 1 week after screening and must have an office msSBP ≥ 145 mmHg and < 180 mmHg after 4 weeks run-in epoch
* patients must successfully complete ABPM and pass technical requirements to be qualified for randomization

Exclusion Criteria:

* Malignant or severe hypertension (grade 3 of WHO classification; msDBP ≥110 mmHg and/or msSBP ≥ 180 mmHg)
* History of angioedema, drug-related or otherwise
* History or evidence of a secondary form of hypertension, including but not limited to any of the following: renal parenchymal hypertension, renovascular hypertension (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease (PKD), drug-induced hypertension
* Patients who previously entered a LCZ696 study and had been randomized or enrolled to receive active drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (21):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fair Oaks, California
  - Novartis Investigative Site, Hawaiian Gardens, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orangevale, California
  - Novartis Investigative Site, Westlake Village, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Conyers, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Richmond, Virginia
- Argentina (6):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires F.D.
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Posadas, Misiones Province
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Philippines (3):
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Quezon City
- Puerto Rico (2):
  - Novartis Investigative Site, Manatí
  - Novartis Investigative Site, Ponce
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
- Spain (6):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Centelles, Catalonia
  - Novartis Investigative Site, Hostalets de Balenya, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alzira, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Started | 188 | 188
Full Analysis Set (FAS) | 188 | 187 (One patient was not included in the SAF and FAS due to mis-randomization.)
Safety Set (SAF) | 188 | 187
Completed | 179 | 175
Not Completed | 9 | 13
Not completed — Adverse Event | 2 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance with study treatment | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Protocol deviation | 3 | 3
Not completed — Subject/guardian decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: Subject demographics and background characteristics by treatment group (Full analysis set)
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg | Total
Number analyzed (Participants) | 188 | 187 | 375
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (10.19) | 58.0 (9.09) | 57.6 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 183
  Male | 97 | 95 | 192

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Mean Ambulatory Systolic Blood Pressure (maSBP)
Description: Twenty-four hour mean ambulatory blood pressure measurements (ABPM) will be performed at baseline and at end of study (week 8). The first 24-hour ABPM will be performed beginning at 24 hours prior to baseline visit and the second will be performed 24 hours prior to week 8 visit.
Time Frame: baseline, 8 weeks
Population: A subset of randomized participants, who had ABPM measurements at both baseline and week 8, were included in the analysis
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 167 | 164
mmHg | -4.26 (0.60) | -1.04 (0.61)
Statistical Analysis 1: Comparison: LCZ696 200 mg vs Olmesartan 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.19, 95% CI 2-sided [-4.73 to -1.65], Standard Error of Mean 0.78

2. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Diastolic Blood Pressure (maDBP)
Description: Twenty-four hour mean ambulatory blood pressure measurements (ABPM) will be performed at baseline and at end of study (week 8). The 24-hour ABPM measurements are performed beginning 24 hours prior to baseline and week 8 visits.
Time Frame: baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 167 | 164
mmHg | -2.27 (0.39) | -0.35 (0.39)

3. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Sitting blood pressure (BP) measurement will be taken at every visit from screening through end of study. For each participant at each visit, four separate sitting BP measurements will be obtained (with a full two minute interval between measurements) and averaged to obtain the mean
Time Frame: baseline, 8 weeks
Population: Full Analysis Set (FAS) - All patients who were randomized. Following the intent to treat principle, patients were analyzed according to the treatment they were assigned to at the randomization. However, patients who were not qualified for randomization and were inadvertently randomized into the study were excluded from the FAS.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
mmHg | -14.21 (1.28) | -10.03 (1.29)

4. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 3
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
mmHg | -7.52 (0.70) | -4.47 (0.71)

5. Secondary Outcome: Change From Baseline in Office Pulse Pressure
Description: Mean sitting pulse pressure (msPP) will be calculated at screening through end of study at every visit. Mean sitting pulse pressure is calculated as msSBP-msDBP.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
mmHg | -6.67 (0.94) | -5.54 (0.94)

6. Secondary Outcome: Number of Patients Achieving Successful Overall Blood Pressure Control
Description: Successful overall blood pressure control is defined as both msSBP/msDBP <140/90 mmHg
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
Participants | 76 | 52

7. Secondary Outcome: Number of Patients Achieving Successful Mean Sitting Systolic Blood Pressure (msSBP) Control
Description: Successful mean sitting systolic blood pressure control is defined as msSBP <140 mmHg
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
Participants | 84 | 58

8. Secondary Outcome: Number of Patients Achieving Successful Mean Sitting Diastolic Blood Pressure (msDBP) Control
Description: Successful mean sitting diastolic blood pressure control is defined as msDBP <90 mmHg
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
Participants | 133 | 112

9. Secondary Outcome: Number of Patients Achieving Successful Mean Sitting Systolic Blood Pressure (msSBP) Response
Description: Successful mean sitting systolic blood pressure response is defined as msSBP <140 mmHg or a reduction ≥ 20 mmHg from baseline.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
Participants | 90 | 65

10. Secondary Outcome: Number of Patients Achieving Successful Mean Sitting Diastolic Blood Pressure (msDBP) Response
Description: Successful mean sitting diastolic blood pressure response is defined as msDBP <90 mmHg or a reduction ≥10 mmHg from baseline.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
Participants | 137 | 115

11. Secondary Outcome: Number of Patients With Total Adverse Events, Serious Adverse Events and Death
Description: Number of patients with total adverse events, serious adverse events and death were reported.
Time Frame: 8 weeks
Population: Safety Set (SAF) - All patients who received at least one dose of study medication in the double-blind epoch. Patients were analyzed according to the treatment they received. One patient was not included in the SAF due to mis-randomization.
Measure: Number; unit: Number of participants
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Number analyzed (Participants) | 188 | 187
Number of participants
  Adverse events (serious and non-serious) | 44 | 41
  Serious Adverse Events | 0 | 2
  Deaths | 0 | 0

ADVERSE EVENTS:
Arm/Group | LCZ696 200 mg | Olmesartan 20 mg
Serious Adverse Events (participants affected / at risk) | 0/188 | 2/187
Other Adverse Events (participants affected / at risk) | 7/188 | 10/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 200 mg (N=188) | Olmesartan 20 mg (N=187)
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 200 mg (N=188) | Olmesartan 20 mg (N=187)
DIZZINESS (Nervous system disorders) | 2 | 4
HEADACHE (Nervous system disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.